CLINICAL TRIAL: NCT03159195
Title: TREATMENT PATTERNS AND CLINICAL OUTCOMES AMONG PATIENTS RECEIVING PALBOCICLIB COMBINATIONS FOR HR+/HER2- ADVANCED/METASTATIC BREAST CANCER IN REAL WORLD SETTINGS
Brief Title: Ibrance Real World Insights
Acronym: IRIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481090; IRIS (Other: Alias Study Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Malignant Neoplasm of Breast
Keywords: metastatic breast cancer; advanced breast cancer; HR+/ HER2-
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR+/HER2- advanced/metastatic breast cancer patients across multiple countries.

SUMMARY:
To describe patient demographics, clinical characteristics, treatment patterns and clinical outcomes of adult female patients who have received palbociclib combination treatments in line with regional licensed indications in real world settings across multiple countries.

ELIGIBILITY:
Physician inclusion criteria

* Oncologist or gynecologist
* Responsible for treating a minimum of ≥2-6 (depending on country) ABC/MBC patients who meet the eligibility criteria.
* Agrees to participate in the study and complete the eCRFs within the data collection period.

Patient inclusion criteria

* Female
* ≥18 years old.
* HR+/HER2- breast cancer diagnosis with confirmed metastatic or advanced disease.
* Received palbociclib plus letrozole/aromatase inhibitor or palbociclib plus fulvestrant in line with the licenced indication(s).
* No prior or current enrolment in an interventional clinical trial for ABC/MBC.
* Minimum of three months of follow up data since palbociclib with fulvestrant initiation, or minimum of six months of follow up data since palbociclib with letrozole/aromatase inhibitor initiation (core medical record review).
* Minimum of three months of follow up data since palbociclib initiation (German interim medical record review only).
* Inoperable or recurrent breast cancer (Japan only)

Exclusion criteria:

Physician exclusion criteria

* Qualified less than 2 years ago or more than 35 years ago
* Participated in observational research for ABC/MBC in the last 3 months
* Have not prescribed either palbociclib plus fulvestrant or palbociclib plus aromatase inhibitor in line with the licenced indication(s).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only
Study Population: Adult female patients with HR+/HER2 advanced or metastatic breast cancer receiving palbociclib combination regimens as per the approved indication.
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Mycock K, Zhan L, Hart K, Taylor-Stokes G, Milligan G, Atkinson C, Mitra D. Real-world treatment patterns and clinical outcomes in patients receiving palbociclib combinations for HR+/HER2- advanced/metastatic breast cancer in Japan: Results from the IRIS study. Cancer Treat Res Commun. 2022;32:100573. doi: 10.1016/j.ctarc.2022.100573. Epub 2022 May 6. PMID 35567914
- [Derived] Mycock K, Zhan L, Taylor-Stokes G, Milligan G, Mitra D. Real-World Palbociclib Use in HR+/HER2- Advanced Breast Cancer in Canada: The IRIS Study. Curr Oncol. 2021 Jan 24;28(1):678-688. doi: 10.3390/curroncol28010066. PMID 33498797
- [Derived] Waller J, Mitra D, Mycock K, Taylor-Stokes G, Milligan G, Zhan L, Iyer S. Real-World Treatment Patterns and Clinical Outcomes in Patients Receiving Palbociclib for Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced or Metastatic Breast Cancer in Argentina: The IRIS Study. J Glob Oncol. 2019 May;5:JGO1800239. doi: 10.1200/JGO.18.00239. PMID 31050919
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481090

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received palbociclib plus aromatase inhibitor (P + AI) or palbociclib plus fulvestrant (P + FV) as treatment of hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) advanced or metastatic breast cancer (ABC/MBC) in April 2017 or later, were observed retrospectively for treatment patterns and clinical outcomes.
Groups:
- Palbociclib + Aromatase Inhibitor (AI) (P+AI): Participants who received palbociclib along with AI for the treatment of ABC/MBC as part of their routine treatment were observed retrospectively for a period of 4 years, approximately.
- Palbociclib + Fulvestrant (P+FV): Participants who received palbociclib along with FV for the treatment of ABC/MBC as part of their routine treatment were observed retrospectively for a period of 4 years, approximately.
Period: Overall Study
Arm/Group | Palbociclib + Aromatase Inhibitor (AI) (P+AI) | Palbociclib + Fulvestrant (P+FV)
Started | 360 | 292
Completed | 360 | 292
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included participants aged >=18 years, diagnosed with HR+/HER- breast cancer with confirmed ABC/MBC, received palbociclib + letrozole/AI or palbociclib + fulvestrant in line with the licensed indication, had no prior or current enrolment in an interventional clinical trial for ABC/MBC, had minimum of 3 months of follow up data since palbociclib with fulvestrant initiation, or minimum of 6 months of follow up data since palbociclib with letrozole/AI initiation.
Groups:
- Palbociclib + Aromatase Inhibitor (P+AI): Participants who received palbociclib along with AI for the treatment of ABC/MBC as part of their routine treatment were observed retrospectively for a period of 4 years, approximately.
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV) | Total
Number analyzed (Participants) | 360 | 292 | 652
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (10.4) | 63.0 (11.4) | 64.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 292 | 652
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: White/Caucasian | 221 | 170 | 391
  Race and Ethnicity: African American | 70 | 49 | 119
  Race and Ethnicity: Asian | 9 | 15 | 24
  Race and Ethnicity: Hispanic/Latino | 40 | 31 | 71
  Race and Ethnicity: Other | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Month 12
Description: PFS was defined as the time from palbociclib combination treatment initiation until 1) clinician documented disease progression (PD) while on palbociclib, 2) death, 3) start of a new therapy line after final palbociclib dose, if the reason for discontinuation of palbociclib was disease progression, or 4) last available follow-up, whichever occurred first. Participants who did not experience a progression event (items 1, 2 and 3) were censored at date of last available follow-up. PFS (in months) was calculated as (first event date - palbociclib initiation date + 1)/30.4. Progressive disease - An increase in visible disease and/or presence of any new lesions; included cases where the clinician indicated progressive disease. Percentage of participants with PFS events at 12 months based on the Kaplan-Meier estimate were reported.
Time Frame: Day 1 of palbociclib combination treatment up to Month 12 (data recorded during 4 years of retrospective observation period)
Population: FAS population included participants aged >=18 years, diagnosed with HR+/HER- breast cancer with confirmed ABC/MBC, received palbociclib + letrozole/AI or palbociclib + fulvestrant in line with the licensed indication, had no prior or current enrolment in an interventional clinical trial for ABC/MBC, had minimum of 3 months of follow up data since palbociclib with fulvestrant initiation, or minimum of 6 months of follow up data since palbociclib with letrozole/AI initiation.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
Number analyzed (Participants) | 360 | 292
Percentage of participants | 84.1 | 79.8

2. Primary Outcome: Percentage of Participants With Progression Free Survival at Month 24
Description: PFS was defined as the time from palbociclib combination treatment initiation until 1) clinician documented disease progression (PD) while on palbociclib, 2) death, 3) start of a new therapy line after final palbociclib dose, if the reason for discontinuation of palbociclib was disease progression, or 4) last available follow-up, whichever occurred first. Participants who did not experience a progression event (items 1, 2 and 3) were censored at date of last available follow-up. PFS (in months) was calculated as (first event date - palbociclib initiation date + 1)/30.4. Progressive disease - An increase in visible disease and/or presence of any new lesions; included cases where the clinician indicated progressive disease. Percentage of participants with PFS events at 24 months based on the Kaplan-Meier estimate were reported.
Time Frame: Day 1 of palbociclib combination treatment up to Month 24 (data recorded during 4 years of retrospective observation period)
Population: FAS population was analyzed for this outcome measure. Data for this outcome measure for reporting group ''P+FV'' was not collected due to limited time on treatment for participants in this group, data was not available beyond Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI)
Number analyzed (Participants) | 360
Percentage of participants | 64.3

3. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) on palbociclib combination therapy according to the RECIST version 1.1 recorded from first dose of study treatment until disease progression due to any cause. Complete response: complete resolution of all visible disease. Partial response: partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: From initiation of treatment up to disease progression (data recorded during 4 years of retrospective observation period)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
Number analyzed (Participants) | 360 | 292
Percentage of participants | 79.5 | 74.0

4. Primary Outcome: Percentage of Participants Alive After 1 Year Post Palbociclib Treatment Initiation
Description: Percentage of participants alive from date of initiation of palbociclib treatment through up to 2 or above progression-based lines of therapy were recorded and reported in this outcome measure. Percentage of participants who alive after 1 year post Palbociclib treatment initiation were based on the Kaplan-Meier estimate.
Time Frame: 1 Year (Month 12) post Palbociclib treatment initiation (data recorded during 4 years of retrospective observation period)
Population: FAS:participants aged >=18 years, diagnosed with HR+/HER- breast cancer with confirmed ABC/MBC, received P + letrozole/AI or P + FV in line with licensed indication, had no prior or current enrolment in an interventional clinical trial for ABC/MBC, had minimum of 3 months of follow up data since P with FV initiation, or minimum of 6 months of follow up data since P with letrozole/AI initiation. "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
Number analyzed (Participants) | 354 | 290
Percentage of participants | 95.1 | 87.9

5. Primary Outcome: Percentage of Participants Alive After 2 Years Post Palbociclib Treatment Initiation
Description: Percentage of participants alive from date of initiation of palbociclib treatment through up to 2 or above progression-based lines of therapy were recorded and reported in this outcome measure. Percentage of participants who alive after 2 years post Palbociclib treatment initiation were based on the Kaplan-Meier estimate.
Time Frame: 2 years (Month 24) post Palbociclib treatment initiation (data recorded during 4 years of retrospective observation period)
Population: FAS population was analyzed for this outcome measure. Data for this outcome measure for reporting group ''P+FV'' was not collected due to limited time on treatment for participants in this group, data was not available beyond Month 12. Here, "Overall Number of Participants Analyzed signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI)
Number analyzed (Participants) | 354
Percentage of participants | 90.1

6. Other Pre Specified Outcome: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who achieved complete (where 'complete response' was recorded at any time on treatment) or partial response (where 'partial response' was recorded at any time on treatment), or stable disease at greater than equal to (>=) 24 weeks on palbociclib combination therapy. Stable disease was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater. Complete response - Complete resolution of all visible disease. Partial response - Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
Number analyzed (Participants) | 360 | 292
Percentage of participants | 93.8 | 93.2

7. Other Pre Specified Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response was defined as the percentage of participants who achieved complete (where 'complete response' was recorded at any time on treatment), partial response (where 'partial response' was recorded at any time on treatment) and stable disease at greater than equal to (>=) 24 weeks on palbociclib combination therapy. Stable disease was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater.
Time Frame: as for outcome 3
Population: FAS population was analyzed. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
Number analyzed (Participants) | 356 | 281
Percentage of participants
  Complete Response | 11.0 | 8.5
  Partial Response | 68.5 | 65.5
  Stable Disease >=24 Weeks | 14.3 | 11.0
  Stable Disease <24 Weeks | 1.4 | 3.2

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected for the study
Description: Due to non-interventional nature of the study, safety data was not collected.
Arm/Group | Palbociclib + Aromatase Inhibitor (P+AI) | Palbociclib + Fulvestrant (P+FV)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT03159195/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03159195/SAP_001.pdf